CLINICAL TRIAL: NCT05228132
Title: A Prospective, Multi-Center, Single-Arm Clinical Study of the Pristine™ Long-Term Hemodialysis Catheter
Brief Title: The Pristine Post-Market Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to considerable changes in the clinical landscape post Covid-19, leading to difficulties executing the study. Results were blinded at time of termination.
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDPI-21-001
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Results first posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-03

CONDITIONS: Kidney Failure, Chronic; Hemodialysis Complication; Hemodialysis Catheter Infection; Hemodialysis Access Failure; Central Venous Catheter Related Bloodstream Infection; End Stage Renal Disease
Keywords: Kidney Replacement Therapy; Hemodialysis; Vascular Access
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pristine™ Long-Term Hemodialysis Catheter (Experimental): The Pristine™ Long-Term Hemodialysis Catheter is a chronic hemodialysis catheter consisting of a dual lumen radiopaque shaft with a pre-formed split tip, which enables long-term vascular access for hemodialysis. The device is intended to be used in patients suffering from chronic kidney disease. The Pristine™ Catheter will be placed according to the Instructions for Use (IFU).
  Interventions: Device: Pristine™ Long-Term Hemodialysis Catheter

INTERVENTIONS:
Device: Pristine™ Long-Term Hemodialysis Catheter — Placement of the Pristine™ Long-Term Hemodialysis Catheter Placement.

SUMMARY:
This is a prospective, multi-center, single-arm study designed to assess the safety and performance of the Pristine™ Long-Term Hemodialysis Catheter.

DETAILED DESCRIPTION:
A total of 142 patients will be enrolled and have the Pristine™ Long-Term Hemodialysis Catheter placed. Under the current enrollment assumptions, up to 15 investigational sites in the United States (US) will participate. Eligible participants will have End Stage Renal Disease requiring hemodialysis through a tunneled dialysis catheter. Follow-up for all enrolled participants will be performed at 1-month, 3-months, 6-months, and 12-months post-Index Procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The participant or legally designated representative must voluntarily sign and date the approved Informed Consent Form (ICF) prior to collection of study-specific data or performance of study-specific procedures.
2. The participant must be willing and able to comply with protocol requirements, including all study visits and procedures.
3. The participant must be either a male or non-pregnant female ≥18 years of age.
4. The participant must have a diagnosis of End Stage Renal Disease with indication for a tunneled dialysis catheter creation.
5. Participant must require chronic hemodialysis treatments 3 times per week with intended use of the Pristine™ Long-Term Hemodialysis Catheter.
6. The participant meets the indications for hemodialysis use and does not meet any of the contraindications per the Pristine Instructions for Use (IFU).
7. The participant must have a patent jugular vein or subclavian vein.

Exclusion Criteria:

1. The participant has known central venous stenosis
2. Based on the local primary investigator's discretion, the patient would not be an appropriate study candidate.
3. The participant has already undergone an AVF or AVG procedure and is awaiting maturation.
4. The participant has an active infection at the time of study enrollment.
5. The participant has a presence of bacteremia or infection within 7 days prior to enrollment.
6. The participant has a history neutropenia or a history of severe immunodeficiency disease.
7. The participant has uncontrolled abnormal coagulation parameters and are at additional risk for clotting or excessive bleeding at time of enrollment per physicians opinion.
8. The participant has a known allergy, intolerance or sensitivity to heparin, or previous incidence of heparin-induced thrombocytopenia.
9. The participant has a known allergy or hypersensitivity to any of the device materials or Ethylene oxide (EtO).
10. The participant has another medical condition or treatment, which in the opinion of the investigator, the participant may be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for completion of study procedures and follow-up.
11. The participant is currently participating in an investigational drug or another device study that has not completed the study treatment or that clinically interferes with the study endpoints. Note: Studies requiring extended follow-up visits for products that were investigational but have since become commercially available, are not considered investigational studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Hoggard, MD, Principal Investigator — Raleigh Access Center
Locations (6):
- United States (6):
  - Trinity Research Group LLC, Dothan, Alabama
  - Yale University, New Haven, Connecticut
  - Louisiana State University Health Shreveport Medical Center, Shreveport, Louisiana
  - Henry Ford Health System, Detroit, Michigan
  - North Carolina Nephrology, PA, Raleigh, North Carolina
  - JML Research Associates, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Started | 7
1-Month Follow-up | 2
3-Month Follow-up | 0
6-Month Follow-up | 0
12-Month Follow-up | 0
Completed | 0
Not Completed | 7
Not completed — Investigation Early Termination by Sponsor | 2
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1
Not completed — Arteriovenous-fistula mature | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Complication Rate of the Pristine™ Catheter
Description: The combined Primary Endpoint is the overall rate of infectious complications and non-infectious complications requiring revision to maintain patency and improve access performance, evaluated against a performance goal (PG) derived from the Dialysis Outcomes and Practice Patterns Study (DOPPS) data.
Time Frame: At 3 months post index procedure.
Population: No participants were followed out to the 3-Month follow-up thus the primary endpoint analysis was not performed. With no source verification or analysis performed, there may be inaccurate reporting and potential misrepresentation of the result.
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Number analyzed (Participants) | 0

2. Secondary Outcome: Rate of Freedom From Catheter-related Bloodstream Infection (CRBSI)
Description: 2019 KDOQI Guidelines for CRBSI defined as, clinical manifestations and at least 1 positive blood culture result from a peripheral source (dialysis circuit or vein) and no other apparent source, with either positive semiquantitative (>15 CFU/catheter segment, hub or tip) or quantitative (>102 CFU/catheter segment, eg, hub or tip) culture, whereby the same organism (species and antibiogram) is isolated from the catheter segment (eg, hub or tip) and a peripheral source (dialysis circuit or vein) blood sample.
Time Frame: 1-month Post-Index Procedure.
Population: No data was collected out to the timepoints following 1-month due to early study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Number analyzed (Participants) | 7
Participants | 6

3. Secondary Outcome: Rate of Freedom From Device and/or Procedure-related Adverse Events
Description: Number of participants free from Device and/or Procedure-related adverse events.
Time Frame: 1-month Post-Index Procedure.
Population: No data was collected out to the timepoints following 1-month due to early study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Number analyzed (Participants) | 7
Participants | 4

4. Secondary Outcome: Rate of Technical Success
Description: Number of Participants with successful placement of the Pristine™ Long-Term Hemodialysis Catheter
Time Frame: At time of Index Procedure.
Population: No data was collected out to the timepoints following 1-month due to early study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Number analyzed (Participants) | 7
Participants | 7

5. Secondary Outcome: Overall Participant Survival Rate
Description: Number of participants that have not died from any catheter related complication.
Time Frame: 1-month Post-Index Procedure.
Population: No data was collected out to the timepoints following 1-month due to early study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Number analyzed (Participants) | 7
Participants | 7

6. Secondary Outcome: Overall Catheter Survival Rate
Description: Number of participants with whom the Pristine™ Catheters have not been removed for any cause.
Time Frame: 1-month Post-Index Procedure
Population: No data was collected out to the timepoints following 1-month due to early study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Number analyzed (Participants) | 7
Participants | 4

7. Secondary Outcome: Overall Patency Rate
Description: Number of participants with their Pristine™ catheter having the ability to achieve a mean dialysis blood flow of ≥300mL/min without need for additional interventions.
Time Frame: 1-month Post-Index Procedure
Population: No data was collected out to the timepoints following 1-month due to early study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Number analyzed (Participants) | 7
Participants | 5

8. Other Pre Specified Outcome: Kit Component Safety and Performance
Description: Defined as the overall rate of the catheter's procedure kit component complications from time of procedure to discharge.
Time Frame: From Index Procedure to Discharge, of which every participant was same day procedure to discharge.
Population: No data was collected out to the timepoints following 1-month due to early study termination.
Measure: Number; unit: Kit Component Complications
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
Number analyzed (Participants) | 7
Kit Component Complications | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Index Procedure to the 1-month Endpoint or until study termination which on average was 42 days, a minimum of 17 days, and a maximum of 77 days.
Arm/Group | Pristine™ Long-Term Hemodialysis Catheter
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pristine™ Long-Term Hemodialysis Catheter (N=7)
Not Device Related-Septic Shock (Infections and infestations) | 1 (1) — Sepsis - bacteraemia, viraemia and fungaemia - Day 17 - Not Related to Device or Procedure
Device Related-Thrombosis in device (Product Issues) | 1 (1) — Thrombosis in device - Clotted Catheter - Day 55 - Likely device related, Unlikely procedure related
Device Related-Thrombosis in device (Product Issues) | 1 (1) — Thrombosis in device - Clotted Catheter - Day 20 - Likely device related, Not procedure related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pristine™ Long-Term Hemodialysis Catheter (N=7)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) — Procedural Pain - Acute Post-Op Pain - Day 0 - Not device related, Likely procedure related
Dizziness (Nervous system disorders) | 1 (1) — Dizziness - Day 40 - Not procedure or device related

LIMITATIONS AND CAVEATS:
Early termination was due to considerable changes in the clinical landscape post Covid-19, leading to difficulties executing the study. Results were not source verified nor study data analyzed prior to termination. Given the sample size no analysis was performed on the limited data available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT05228132/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT05228132/SAP_001.pdf